CLINICAL TRIAL: NCT06444061
Title: Cultural Adaptation and Psychometric Validation of the Balance Recovery Confidence Scale (BRCS) in Older Turkish Adults
Brief Title: The Balance Recovery Confidence (Brc) Scale
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Abdulkadir dağbaşı, Principal Investigator, Necmettin Erbakan University
Other Study IDs: ADagbasi003
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Accidental Falls; Balance; Distorted; Aging; Self Efficacy; Adaptation, Psychological
Keywords: Balance confidence; fall risk; cultural adaptation; geriatrics; psychometric properties

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cross-sectional study is to evaluate the cultural adaptation, reliability, and validity of the Turkish version of the Balance Recovery Confidence Scale (BRCS), named Dengeyi Düzeltmede Kendine Güven Ölçeği (DDKGÖ), in older Turkish adults aged 65 and above. The main questions it aims to answer are:

Does the Turkish adaptation (DDKGÖ) demonstrate acceptable cultural validity, internal consistency, and test-retest reliability in measuring balance recovery confidence?

How does the DDKGÖ correlate with established tools assessing fear of falling, balance confidence, and physical performance (e.g., FES-I, ABC, TUG) to confirm convergent validity?

Participants will:

Complete the DDKGÖ questionnaire twice (7 days apart) to assess test-retest reliability.

Undergo physical performance tests (e.g., Timed Up and Go, Handgrip Strength Test, 30-Second Chair Stand Test).

Provide responses to additional self-report scales (FES-I, ABC) to evaluate convergent validity.

This study focuses on community-dwelling older adults without severe cognitive or physical impairments. Results will help standardize the DDKGÖ as a tool for identifying fall risk and personalizing rehabilitation strategies in Turkish geriatric populations.

DETAILED DESCRIPTION:
This observational psychometric study is designed to establish the cultural validity, reliability, and overall measurement performance of the Turkish adaptation of the Balance Recovery Confidence Scale (DDKGÖ) in community-dwelling older adults. After obtaining informed consent and confirming basic eligibility, participants will undergo a two-phase assessment protocol with a one-week interval between phases.

During Phase 1, each participant will complete a structured interview and self-report questionnaires in a single session. These include the 19-item DDKGÖ (to assess reactive balance confidence), the Falls Efficacy Scale-International, and the Activities-specific Balance Confidence Scale. Trained assessors will also record demographic and health information (e.g., age, sex, comorbidities, history of falls) and administer a battery of standardized performance tests-such as the Timed Up and Go, 30-Second Chair Stand, Tinetti Balance & Gait, and Handgrip Strength tests-to evaluate convergent validity.

Exactly seven days later, in Phase 2, participants will return to repeat the DDKGÖ under identical conditions to evaluate test-retest stability. All sessions will be conducted in the same clinical setting by the same examiners, using standardized instructions and order of administration to minimize procedural variability.

Collected data will be anonymized and entered into a secure database. Statistical analyses will include exploratory and confirmatory factor analyses to examine structural validity, calculation of internal consistency (e.g., Cronbach's α), intraclass correlation coefficients for test-retest reliability, Bland-Altman limits of agreement to quantify measurement error, and correlation analyses with existing balance- and fear-of-fall measures and performance tests to establish convergent validity.

By following this stepwise process-translation verification, initial validity and reliability testing, and retest assessment-this study will provide a comprehensive evaluation of whether the DDKGÖ is suitable for use in both research and clinical practice to identify older Turkish adults at elevated fall risk and to monitor changes in their confidence to recover from postural disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years.
* Community-dwelling individuals capable of independent living (use of walking aids permitted).
* Literate in Turkish.
* Ability to complete 6 meters of walking within 12 seconds.
* Ability to grasp a 30 cm ruler with both hands.

Exclusion Criteria:

* Requiring assisted mobility outside the home.
* Mini-Mental State Examination (MMSE) score ≤23.
* Timed Up and Go (TUG) test duration >12 seconds.
* Active malignancy or history of myocardial infarction/cardiac surgery within the last 3 months.
* Structural heart disease, severe COPD, or oxygen dependence.
* Musculoskeletal/neurologic disorders affecting balance or muscle function (e.g., Parkinson's disease, stroke sequelae, multiple sclerosis, severe dementia, epilepsy).
* Fracture within the last 6 months.
* Vision or hearing loss impairing assessment participation.
* Inability to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population will consist of community-dwelling older adults aged 65 years and older, recruited from a single center in Turkey. Participants must be literate in Turkish, capable of independent living (with or without walking aids), and able to perform basic mobility tasks such as walking 6 meters within 12 seconds. Exclusion criteria will include cognitive impairment (MMSE ≤23), mobility limitations (Timed Up and Go >12 seconds), recent fractures (within the last 6 months), severe cardiopulmonary or neurological conditions, and significant sensory impairments. Educational background, fall history, and sociodemographic characteristics will be documented to describe the sample.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Balance Recovery Confidence Scale (BRCS) | Start (initial assessment session, Day 1) and 7 days later (follow-up session on Day 8)
  The BRCS is a 19-item self-report scale developed to assess individuals' perception of self-efficacy for the restoration of balance after postural perturbations (such as stumbling, slipping, sudden loss of balance).

SECONDARY OUTCOMES:
Falls Efficacy Scale-International ( FES-I ) | Baseline administration (Day 1)
  The FES-I is a valid and reliable self-report scale consisting of 16 items designed to assess the subjective level of concern about the fear of falling during activities of daily living.
Activities-specific Balance Confidence Scale ( ABC ) | Baseline administration (Day 1)
  The ABC is a sixteen-item self-report tool that subjectively assesses individuals' confidence levels in maintaining balance during activities of daily living.
Timed Up and Go ( TUG ) | Baseline administration (Day 1)
  The TUG is a standardized clinical performance measurement protocol developed to measure the functional mobility capacity of individuals, assessing dynamic postural control, gait kinematics and movement strategies during activity transitions.
Handgrip Strength Test ( HGST ) | Baseline administration (Day 1)
  HGST is an objective neuromuscular assessment method used to quantitatively measure the maximal isometric contraction capacity of the hand and forearm muscles.
Tinetti Balance & Gait Test ( TBT&TGT ) | Baseline administration (Day 1)
  TBT&TGT is a 16-item performance scale developed to clinically analyze postural stability, ambulation skills and dynamic balance control in elderly individuals.
30-Second Chair Stand Test ( 30s-CST ) | Baseline administration (Day 1)
  The 30s-CST is a widely used functional measurement tool for assessing lower extremity muscle endurance and dynamic balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: abdulkadir dağbaşı, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soh SL, Tan CW, Xu T, Yeh TT, Bte Abdul Rahman F, Soon B, Gleeson N, Lane J. The Balance Recovery Confidence (BRC) Scale. Physiother Theory Pract. 2024 Mar 3;40(3):658-669. doi: 10.1080/09593985.2022.2135420. Epub 2022 Oct 19. PMID 36259660